CLINICAL TRIAL: NCT02959021
Title: Primary Care Obesity Management in the Southeast_PROMISE
Brief Title: Partnership Optimizes Weight Management in Primary Care
Acronym: PROMISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gareth R. Dutton PhD, Associate Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIH R01DK106041; R01DK106041 (NIH)
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obesity
Keywords: weight loss; behavioral; primary care; lifestyle
MeSH Terms: conditions — Obesity; Weight Loss; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-directed treatment (Active Comparator): Participants randomly assigned to this arm will receive written and pre-recorded behavioral weight loss intervention materials (i.e., DVDs, online videos), and they will be instructed to work through the materials independently at their own pace. They will have continued physician contact as needed for routine medical care.
  Interventions: Behavioral: weight loss intervention - self directed
- Peer coach treatment (Experimental): Participants randomly assigned to this arm will receive a combination of in-person, group-based behavioral weight loss sessions plus individual, telephone contacts. Groups and phone calls will be facilitated by a peer coach interventionist. Similar to the self-directed condition, participants will receive written and pre-recorded intervention materials (i.e., DVDs, online videos). They will also have continued contact with their physician for routine medical care.
  Interventions: Behavioral: weight loss intervention - peer coach

INTERVENTIONS:
Behavioral: weight loss intervention - self directed
  Arms: Self-directed treatment
Behavioral: weight loss intervention - peer coach
  Arms: Peer coach treatment

SUMMARY:
The purpose of this study is to examine whether a primary care weight management intervention delivered by peer coaches produces greater weight loss than a self-directed program without peer coach support.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-75 years
* Body mass index (BMI) 30-50 kg/m2
* Receiving primary care services at one of the practices participating in this study

Exclusion Criteria:

* Uncontrolled hypertension (blood pressure >160/100 mm Hg at screening)
* Any of the following other medical conditions: myocardial infarction or cerebrovascular accident within the last six months; unstable angina within the past six months; NYHA Class III or IV congestive heart failure; type 1 diabetes; cancer requiring treatment in past five years (exception: non-melanoma skin cancer); and chronic lung diseases that limit physical activity
* Current use of any of the following medications: antipsychotic agents, monoamine oxidase inhibitors, systemic corticosteroids, or chemotherapeutic drugs; prescription weight loss medications (past six months)
* Unwilling or unable to do any of the following: give informed consent; read/understand English; accept random assignment; travel to the intervention site
* Likely to relocate out of the area in the next 2 years
* Participation in another randomized research project
* Weight loss > 10 pounds in past six months
* History of bariatric surgery

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
body weight | 6, 12, and 18 months
  change in body weight (kg) from baseline to follow-up assessments

SECONDARY OUTCOMES:
physical activity | 6, 12, and 18 months
  Self-reported physical activity assessed via the Paffenbarger Physical Activity Questionnaire (PPAQ).
treatment adherence | 6, 12, and 18 months
  Treatment adherence will be assessed by the number of treatment sessions and phone calls completed.
treatment burden | 6, 12, and 18 months
  Behavioral burden of treatment will be assessed with self-report questionnaires including items about the perceived burden of behavioral targets such as self-monitoring, dietary changes, maintaining physical activity, and the impact of treatment on social relationships.
treatment satisfaction | 6, 12, and 18 months
  Participants will complete self-report items assessing their attitudes and satisfaction regarding the weight loss intervention and weight loss achieved.
side effects | 6, 12, and 18 months
  Symptom checklist including minor (e.g., constipation, dry mouth) and more severe events (e.g., cardiovascular events) will be administered to assess potential adverse side effects associated with treatment.
quality of life | 6, 12, and 18 months
  Quality of life will be assessed through the validated Short-Form 12 (SF-12), which provides measures of health-related quality of life for physical and mental health.
physical and social functioning | 6, 12, and 18 months
  Items from the Patient Reported Outcome Measurement Information System (PROMIS) will be administered, including the 8-item short forms for physical and social functioning.
mood | 6, 12, and 18 months
  The Patient Health Questionnaire-8 (PHQ-8), a validated self-report measure of depressive symptoms experienced over the past two weeks, will be administered.
healthcare utilization | 6, 12, and 18 months
  Self-reported utilization of health care services (hospitalizations, ER/physician office visits, prescription drugs, etc.) and out-of-pocket costs will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Dutton, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
With the documented permission of the IRB, the PI may develop a transportable de-identified database, codebook, and mechanism by which data can be shared with qualified investigators. Interested investigators will be asked to complete a standardized request form stating the specific aims of the analyses, the analytic plan, available resources for completing the proposed project, proposed timeline, and goals (i.e., manuscripts, presentations, and/or grant applications). The PI and research team will review these requests to determine whether the proposed analyses constitute an innovative and significant exploration of the data, whether the proposed team has sufficient resources to complete the request, and whether data will be adequately protected and managed. If any of these issues are problematic, the PI and research team will attempt to negotiate a fair resolution with the interested investigators and NIH program staff.

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT02959021/SAP_000.pdf